CLINICAL TRIAL: NCT01228422
Title: Study of Pharmacokinetics and Pharmacodynamics of Alpha Interferon-2A of Blausiegel Trade and Industry the Compared the Product Roferon A, of Laboratory of Roche
Brief Title: Pharmacokinetics and Pharmacodynamics of Interferon Alpha 2A
Acronym: interferon
Status: Completed | Type: Observational
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Other Study IDs: INT2ABLA0908
Record Dates: First submitted 2008-10-21; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Will be studied 24 subjects divided Research and 2 parallel groups; The treatment is a dose of 3MUI of alpha interferon 2nd; There will be collection of blood at times: 0, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours.; The volunteers will be hospitalized 24 hours.; Will be measured labels the AUC, Tmax, Cmax, neopterin and beta2-microglobulin
MeSH Terms: interventions — Interferon alpha-2

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: test interferon - blausiegel
  Interventions: Biological: Interferon alpha 2a
- 2: reference interferon - Roferon A (Roche)
  Interventions: Biological: Interferon alpha 2a

INTERVENTIONS:
Biological: Interferon alpha 2a — 3MUI

SUMMARY:
The aim was to verify the Pharmacokinetics and Pharmacodynamics of alpha interferon product-2A - Blausiegel, taking as the comparator drug product Roferon ® A (interferon alpha-2A - Roche Laboratory).

DETAILED DESCRIPTION:
The Interferons (IFNs) are a group of cytokines produced by vertebrates in response to various stimuli, including the presence of foreign nucleic acids in the body, bacteria, tumor cells and viral antigens. These proteins have significant shares immunomodulatory, antiproliferative and antiviral drugs, the first line of defense of the body. Once produced, the IFNs block viral replication, maximize the lytic activity of natural killer cells, increase the expression of MHC class I in cells infected by viruses and induce the development of Th1 cells The production of interferon alpha-2A is now held by biotechnology with the establishment of a chain of DNA producer of interferon alpha-2a in the chain of original DNA of a bacterium, allowing the bacteria produce this drug on an industrial scale. In the process of synthesis, the 165 amino acids that are part of this molecule can change in your order with no reduction in activity or changes in the properties.

Due to this fact, the biological and medicinal considered, especially those in manufacturing by genetic engineering, need to prove their clinical activity so that they can be marketed. In the case of interferon, the consequences of the use of a product without activity compared to treat patients with Hepatitis C can lead to serious health complications from them. It is therefore necessary to prove its clinical activity and pharmacokinetics before its clinical efficacy. The sponsor of this study aims to end the renewal of registration of interferon alpha-2A with the Ministry of Health So this study to evaluate the Pharmacokinetics and Pharmacodynamics of interferon alpha-2a may allow in the future this medicine can be used by a year in patients with hepatitis C, without risk to their health, besides those already known and inherent in the treatment of any interferon.

ELIGIBILITY:
Inclusion Criteria:

* Accepting the End of Free and Informed Consent;
* Research subjects were male, aged 18 to 55 years;
* Research subjects with body mass index ≥ 19 and ≤ 30;
* Be considered healthy, from the analysis of medical history, medical examination and laboratory tests within the normal range.

Exclusion Criteria:

* Results of laboratory tests outside the values considered acceptable in accordance with the criteria of medical evaluator;
* Having participated in any experimental study or have ingested any experimental drug in the last three months before the start of the study;
* Have made regular use of medication in the past 4 weeks preceding the start of the study or have made use of any medication a week before the start of the study;
* Have been hospitalized for any reason, up to 8 weeks before the start of the study;
* Present history of abuse of alcohol, drugs or medications, or have ingested alcohol within 48 hours prior to the period of stay;
* Have a history of liver disease, renal, pulmonary, gastrointestinal, hematological or psychiatric;
* Present pressure changes of any cause that requires pharmacological treatment; present history of myocardial infarction, angina and / or heart failure;
* Have donated or lost 450 ml of blood or more in the three months preceding the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evaluate in parallel pharmacodynamic parameters and pharmacokinetics. | 96 hours.
  Pharmacokinetic parameters of the drug will be held 17 blood samples over a period of 96 hours. The parameters Cmax, Tmax, area under the curve (AUC), among others, will be quantified in each individual. The pharmacodynamics will be studied from the alteration of endogenous biomarkers sensitive to stimulation by interferon.

SECONDARY OUTCOMES:
Evaluation of clinical safety through a comparison of clinical and laboratory parameters pre-and post-study and the incidence of adverse events | 96 hours.
  The pharmacokinetic parameters of the drug will be held 17 blood samples over a period of 96 hours. The parameters Cmax, Tmax, area under the curve (AUC), among others, will be quantified in each individual. The pharmacodynamics will be studied from the alteration of endogenous biomarkers sensitive to stimulation by interferon.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Doctor, Principal Investigator — Azidus Brasil
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil